CLINICAL TRIAL: NCT02886689
Title: C.O.R.P.U.S. : Observational Cohort of Active Rheumatoid Arthritis, Spondylarthropathy and Idiopathic Juvenile Arthritis in France
Brief Title: C.O.R.P.U.S.: Observational Cohort of Adult and Child Inflammatory Arthritis in France
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GUILLEMIN Francis, MD, Professor, Central Hospital, Nancy, France
Other Study IDs: PCv1.6-12-11-05
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Arthitis, Juvenile Idiopathic
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: patients will be those receiving any biotherapy
  Interventions: Drug: TNF-alpha antagonist and other biotherapy
- 2: patients will be those not receiving biotherapy : non indication, refusal, contraindication.

INTERVENTIONS:
Drug: TNF-alpha antagonist and other biotherapy
  Groups: 1

SUMMARY:
C.O.R.P.U.S. is the first French observatory of care practices in active inflammatory rheumatism of children and adults: rheumatoid arthritis, spondylarthropathy, and idiopathic juvenile arthritis, established under the auspices of national health authorities.

Its goal is to document safety, effectiveness in routine practice of various therapy, including biotherapy, of prescription or non-prescription over 5 years.

A cohort will be constituted including any new case of active disease (DAS 28 > 3,2, BASDAI > 4, failure of methotrexate), without previous prescription of biotherapy. Therefore, it will be possible to have patients non exposed to biotherapy (non indication, refusal, contraindication) compared to patients exposed to biotherapy, and to monitor adverse events occurrence as well as effectiveness in routine practice over time, according to prescription, maintenance or switch of various therapies.

DETAILED DESCRIPTION:
Rational:

Biotherapies, including anti-TNF alpha have demonstrated effectiveness by several randomized clinical trials. The long-term use in clinical practice raise several questions regarding their safety, the risk-benefit ratio, and the actual advantage of such treatment in real life routine practice. Moreover such practice may considerably change, as far as increasing number of therapies are made available on the market.

On request form national health authorities in France, this phase 4 study will help monitor the changing strategies of prescription, the effectiveness and safety of these drugs.

Objectives :

1. to determine the impact of biotherapy prescription in 3 category of diseases assessed on articular, functional and quality of life outcomes, as well as other drug consumption, and to monitor adverse events
2. to determine the place of biotherapy in the sequence of treatments of patients

Study design:

an open cohort study to include patients over 3 years continuously, and to last at least 5 years form study start, with annual prospective follow-up. C.O.R.P.U.S. will be the first French observatory of prescription (or non-prescription) practices of biotherapy in first or switch treatment.

Sample:

Patients will be recruited by French network of private rheumatologist, and 40 university hospital rheumatology ward.

Data collected:

Socio-demographic, clinical parameters, function and quality of life know to have prognostic value

* Exposed patients will be those receiving any biotherapy
* Non-exposed patients will be those not receiving biotherapy : non indication, refusal, contraindication.

Outcomes:

radiographic joint lesions, function, adverse events, maintenance rate, drug consumption.

Sample size:

a sample of 1200 RA, 350 SPA and 300 IJA will be recruited every year for the first 3 years.

Adverse events:

Any adverse events will be reported to the national centre for pharmacovigilance.

IRB:

this protocol has been accepted by the CCTIRS and the CNIL.

Study monitoring:

A scientific committee has been constituted and is in charge of respect of any aspects of the protocol, particularly regarding safety A steering committee has been constituted and includes any drug company representative marketing such therapy, as well as representative of Inserm.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis by rheumatologist of rheumatoid arthritis

* DAS score > 3.2,
* any age of onset
* hand and feet x-ray within the past 3 months
* never received any biotherapy Diagnosis by rheumatologist of spondylarthropathy (ankylosing spondylitis, psoriasic arthritis)
* active disease
* hand and feet (peripheral) or spine (axial) x-ray within the past 3 months Diagnosis by rheumatologist of idiopathic juvenile arthritis
* failure or intolerance to methotrexate
* x-ray within the past 3 months

Exclusion Criteria:

* received previous biotherapy
* other spondylarthropathy than ankylosing spondylitis, psoriasic arthritis

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering rheumatoid arthritis, spondyloarthropathy or idiopathic juvenile arthritis, recruited with rheumatologist in public and private practice
Sampling Method: Non-Probability Sample
Enrollment: 5400 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Drug consumption | first year

CONTACTS AND LOCATIONS:
Overall Officials: Francis Guillemin, MD, PhD, Study Chair — Central Hospital, Nancy, France; Jacques Benichou, MD, PhD, Principal Investigator — CHU, Rouen, France; Alain Sasraux, MD, PhD, Principal Investigator — CHU de la Cavale Blanche, Brest, France; Loic Guillevin, MD, PhD, Principal Investigator — Hopital Cochin, Paris, France; Jean Sibilia, MD, PhD, Principal Investigator — CHU Hautepierre, Strasbourg, France; Anne Marie Prieur, MD, PhD, Principal Investigator — Hopital Necker, Paris , France; Daniel Wendling, MD, PhD, Principal Investigator — CHU Minioz, Besançon, France
Locations (1):
- Central Hospital, Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
open to partnership